CLINICAL TRIAL: NCT00016029
Title: Prospective Comparison of Air Contrast Barium Enema (ACBE), Computed Tomographic Colonography (Virtual Colonoscopy) and Colonoscopy for Evaluation of the Colon in Patients With Fecal Occult Blood
Brief Title: Comparison of Barium Enema, Computed Tomographic Colonography, and Colonoscopy in Detecting Colon Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: 0866; DUMC-000866-00-5R; DUMC-CA14326; NCI-V01-1655; CDR0000068587 (Other: NCI)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2003-09

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Barium Enema

INTERVENTIONS:
Other: screening questionnaire administration
Procedure: barium enema injection
Procedure: computed tomography
Procedure: computed tomography colonography
Procedure: diagnostic colonoscopy
Procedure: screening colonoscopy

SUMMARY:
RATIONALE: Screening tests may help doctors detect cancer cells early and plan more effective treatment for cancer. New diagnostic procedures such as computed tomographic colonography may provide a less invasive method of identifying patients who have colon cancer.

PURPOSE: Diagnostic and screening trial to compare the effectiveness of barium enema, computed tomographic colonography, and colonoscopy in detecting of colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the accuracy of air contrast barium enema, computed tomographic colonography (virtual colonoscopy), and colonoscopy for the detection of colonic lesions in patients with factors related to colon cancer.
* Compare the patient experience during each of these imaging tests.

OUTLINE: This is a multicenter study.

A repeat fecal occult blood test is performed. Patients then undergo an air contrast barium enema (ACBE). At 7-10 days after ACBE, patients undergo a computed tomographic colonography (virtual colonoscopy) followed by a colonoscopy on the same day.

A repeat ACBE may be performed if there is a discrepancy between the initial ACBE and colonoscopy. If the repeat ACBE continues to show an abnormality, patients undergo a second colonoscopy.

Within 24 hours of completion of each test, patients fill out a questionnaire about their experience. At 5-7 days after completion of all tests, patients complete a final questionnaire comparing all 3 tests.

PROJECTED ACCRUAL: A total of 2,133 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following must be present:

  * At least 1 positive fecal occult blood test within the past 6 months
  * Iron deficiency anemia, defined as:

    * Hemoglobin less than 13 g/dL (males)
    * Hemoglobin less than 12 g/dL (females)
    * Ferritin less than 45 g/dL
  * Episode of bright red blood per the rectum
  * Family history of colon cancer or adenoma

    * One first-degree relative diagnosed with colon cancer or adenoma at age 60 or under OR
    * Two first-degree relatives diagnosed with colon cancer or adenoma at any age
* No active gastrointestinal hemorrhage, including any of the following:

  * Reported or witnessed hematemesis
  * Melenic stools
  * Melenemesis
  * Multiple episodes of hematochezia within the past 2 months

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No myocardial infarction or cerebrovascular accident within the past 6 weeks

Pulmonary:

* No respiratory failure within the past 6 weeks

Other:

* No serious medical disorder (e.g., sepsis) within the past 6 weeks
* Weight less than 300 pounds
* Willing and able to undergo endoscopic or radiologic procedures

  * No need for special precautions in performing endoscopic procedures (e.g., antibiotic prophylaxis or complicated anticoagulation reversal)
* No prisoners
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent clinical trial participation involving drugs, medical devices, and/or biologics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2000-08; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Rockey, MD, Study Chair — Duke Cancer Institute
Locations (14):
- United States (14):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - California Pacific Medical Center - Pacific Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Indian River Radiology, Vero Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Troy Internal Medicine, P.C., Troy, Michigan
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Massey Cancer Center, Richmond, Virginia